ID: HF-22003

Title:The Effect of the Mobile Application Developed for the Care of Sick Newborns

NCT Number: NCT05776615

Document Date: June 12, 2024 (IRB approval date)

## **Study Protocol**

Development of Mobile Application

Pre test

Identification of nurses eligible for inclusion in the study

Randomized

Mobile aplication group (n= 31 )

Control grup (n=32 )

Informing nurses about mobile application and research, obtaining written consent from nurses

### Mobile Application group data collection

Collection of Mobile Application Data: The nurses included in the study group filled out the data collection tools (Nurse Descriptive Characteristics form, nursing diagnoses perception scale, 'MISSCARE nursing Determination Questionnaire in the Neonatal Intensive Care Unit) before the application was installed on their phones, the mobile application was introduced, the application was downloaded from Google Play Store or App Store, and how to use the application was explained. Nurses clicked the notifications from the mobile application. In addition, they were asked to prepare and record a care plan using the mobile application from a patient newborn that they care for every week. At the end of the 1st and 3rd months, Nursing Diagnosis Perception Scale, MISSCARE Nursing Questionnaire in the Neonatal Intensive Care Unit, and System Applicability Scale (SUS-TR) were administered to the nurses.

## **Collection of Control Group Data**

The nurses included in the control group were administered the Nurse Descriptive Characteristics form, nursing diagnoses perception scale, 'MISSCARE nursing Determination Questionnaire in the Neonatal Intensive Care Unit. At the end of the 1st and 3rd months, the nursing diagnoses perception scale and the 'MISSCARE nursing Determination Questionnaire in the Neonatal Intensive Care Unit were applied to the nurses. System Applicability Scale (SUSTR) was not applied.

ANALYSING THE DATA AND REPORTING THE RESEARCH

## **Statistical Analysis Plan**

Statistical analysis of the data was performed using SPSS (IBM SPSS Statistics 27) package programme. Frequency tables and descriptive statistics were used to interpret the findings of the study. The conformity of the measurements to normal distribution was analysed using Shapiro-Wilk analysis. Consistent with parametric methods, 'Independent sample t test' was used to compare the measurements of two independent groups. The Repeated Measures (F-table value) method was used to compare the measurements of three or more dependent groups. 'Bonferroni' correction was applied for pairwise comparisons of three or more groups. Nonparametric methods were used for measurements that did not fit the normal distribution. Consistent with nonparametric methods, the 'Mann-Whitney U' test (Z-table value) was used to compare the measurements of two independent groups. The Wilcoxon signed-rank test (Ztable value) was used to compare the measurements of two dependent groups. 'Friedman' test ( $\chi$ 2-table value) was used to compare the measurements of three or more dependent groups. 'Bonferroni' correction was applied for pairwise comparisons of three or more groups. The relationship between two qualitative variables was analysed by Pearson-γ2 cross-tabulations. Spearman's correlation coefficient was used to examine the relationship between two quantitative variables that were not normally distributed. Biostatistics expert support was obtained in the analysis of the data.



Turkish Republic

### AYDIN ADNAN MENDERES UNIVERSITY RECTORATE

# PES Tisolin Consumitation victorical real

Directorate of the Institute of Health Sciences

Non-Interventional Research Ethics Committee

Number: E-21347915-050.04-549014

June 24, 2024

Subject: Regarding your Ethics Committee Application

No. 2022/021.

Associate Professor Dr. Seher SARIKAYA KARABUDAK Faculty Member

Below is the decision number I regarding your study taken at the regular meeting of the Health Sciences Institute Non-Interventional Research Ethics Committee held on June 12, 2024. I present it for your information.

**DECISION: 1** 

Protocol No: 2022/021

Responsible Executive: Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK

The petition of Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK, regarding the final report of her research titled "The Effect of the Mobile Application Developed for the Care of Sick Newborns on Nurses' Perception of Nursing Diagnoses and Unmet Care: A Randomized Controlled Experimental Study", which was approved by the Non-Interventional Research **Ethics** Committee of Aydÿn Adnan Menderes University Health Sciences Institute on 10.06.2022, was discussed on **12.06.2024**.

The petition stated that the study had been completed, and the final report was attached. It was concluded that the study had been conducted and completed within ethical guidelines, and that the requested documents were complete. It was unanimously decided that the study should receive **Ethics Committee Approval**.

Prof. Dr. Turhan DOST

Chairman of the Board

This document has been signed with a secure electronic signature.

Verification Code: BSRA1LTPE9 Central

Verification Address: https://turkiye.gov.tr/ebd?eK=5740&eD=BSRA1LTPE9&eS=549014



## INFORMED CONSENT FORM

# (Control Group)

The study titled "The Effect of the Mobile Application Developed for the Care of Hospitalized Newborns on Nurses' Perception of Nursing Diagnoses and Miss Care: A Randomized Controlled Experimental Study" will be conducted by Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK and Lecturer Canan Sümeyra GÜN.

This randomized controlled experimental study has been designed to determine the effect of the mobile application developed for the care of hospitalized newborns in the Neonatal Intensive Care Unit (NICU) on nurses' perceptions of nursing diagnoses and unmet care, as well as to evaluate the usability of the mobile application. Participation in this study is voluntary. You may choose not to participate or may withdraw while filling out the questionnaires. Data collected through the questionnaires will be used for scientific purposes only. No adverse effects are expected from participating in this study.

During the study, you will be asked to complete the following:

- Nurse Descriptive Characteristics Form (19 items, including age, gender, work experience, etc.),
- Nursing Diagnoses Perception Scale (26 items),
- NICU "Unmet Nursing Care" Questionnaire (69 items).

Completing these forms will take approximately 20–30 minutes. Afterwards, at the end of the 1st month and at the end of the 3rd month, you will again be asked to complete the Nursing Diagnoses Perception Scale (26 items) and the NICU "Unmet Nursing Care" Questionnaire (69 items).

All questions related to the study will be answered by the researchers, Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK and Lecturer Canan Sümeyra GÜN. At the end of the study, if you wish, the mobile application can also be installed on your device for your use.

For any questions related to this study, you may contact:

- Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK at 0505 448 37 03 or ssarikaya@adu.edu.tr
- Lecturer Canan Sümeyra GÜN at 0545 812 57 20 or canansumeyra.gun@ksbu.edu.tr

You may ask during or after the application, either via e-mail or by phone (mobile).

We thank you for your participation.

I, the undersigned, agree to participate in the study titled "The Effect of the Mobile Application Developed for the Care of Hospitalized Newborns on Nurses' Perception of Nursing Diagnoses and Unmet Care: A Randomized Controlled Experimental Study."

Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK and Lecturer Canan Sümeyra GÜN have

Signature:

provided me with detailed verbal and/or written information about the structure, purpose, and possible duration of the study, what is expected from me, and what to do in case of an adverse situation.

I have had the opportunity to ask all questions I had regarding the study to the researchers, and I understood the answers and the information provided to me. I permit Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK and Lecturer Canan Sümeyra GÜN to conduct this study with me, under the condition that they explain the details clearly and maintain the confidentiality of my personal information.

I agree to comply with all the rules throughout the study, to fully cooperate with the researchers, and to contact them immediately if any issue arises. I accept that the results of this study may be used without restriction in publications, reports, or other scientific documents. I also understand that I can withdraw from this study at any time

**Participant** Researcher Name-Surname: Title, Name-Surname: Lecturer Canan Date: Sümeyra Gün/Assoc. Prof. Dr. Seher **SARIKAYA KARABUDAK** Phone No: Date: Signature: Phone No: 05458125729/0505 448 37 03 Signature: **Participant** Name-Surname: Address: Aydın Adnan Menderes University, Central Campus, Faculty of Date: Nursing, Aydın 09100 Phone No:

### INFORMED CONSENT FORM

(Study Group)

The study titled "The Effect of the Mobile Application Developed for the Care of Hospitalized Newborns on Nurses' Perception of Nursing Diagnoses and Miss Care: A Randomized Controlled Experimental Study" will be conducted by Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK and Lecturer Canan Sümeyra GÜN. This randomized controlled experimental study has been designed to determine the effect of the mobile application developed for the care of hospitalized newborns in the Neonatal Intensive Care Unit (NICU) on nurses' perceptions of nursing diagnoses and miss care, as well as to evaluate the usability of the mobile application. Participation in this study is voluntary. You may choose not to participate or may withdraw while filling out the questionnaires. Data collected through the questionnaires will be used only for scientific purposes. No adverse effects are expected from participating in this study. During the study, you will be asked to complete: - Nurse Descriptive Characteristics Form (19 items, such as age, gender, work experience, etc.), - Nursing Diagnoses Perception Scale (26 items), - NICU "MISSCARE" Questionnaire (69 items). Completing these forms will take approximately 30-40 minutes. Afterwards, the mobile application developed for the care of hospitalized newborns will be installed on your phone. You will be provided with a username and password to log in, its functionality will be checked, and you will be informed about its use. During the usage period, you will receive periodic notifications via the mobile application, and you will need to respond by selecting "Yes" or "No." Paying attention to these notifications is important and valuable for the effectiveness of the study. In addition, it is your legal responsibility not to share the mobile application and its content with other nurses. Maintaining this confidentiality during the study is essential for the reliability and accuracy of the results. We kindly ask for your diligence regarding this matter. At the end of the study, this mobile application will also be installed for other nurses upon their request. All questions related to the study and the mobile application will be answered by the researchers, Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK and Lecturer Canan Sümeyra GÜN.

At the end of the 1st month and at the end of the 3rd month after you start using the mobile application, you will again be asked to complete the Nursing Diagnoses Perception Scale (26 items), the NICU "MISSCARE" Questionnaire (69 items), and the System Usability Scale (10 items). For any questions related to this research, you may contact: - Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK at 0505 448 37 03 or ssarikaya@adu.edu.tr - Lecturer Canan Sümeyra GÜN at 0545 812 57 20 or canansumeyra.gun@ksbu.edu.tr You may ask during or after the application, either via e-mail or by mobile phone. We thank you for your participation.

I, the undersigned, agree to participate in the study titled "The Effect of the Mobile Application Developed for the Care of Hospitalized Newborns on Nurses' Perception of Nursing Diagnoses and Miss Care: A Randomized Controlled Experimental Study." Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK and Lecturer Canan Sümeyra GÜN have provided me with detailed verbal and/or written information about the structure, purpose, and possible duration of the study, what is expected from me, and what to do in case of an adverse situation. I have had the opportunity to ask all questions I had regarding the study to the researchers, and I understood the answers and the information provided to me. I permit Assoc. Prof. Dr. Seher SARIKAYA KARABUDAK and Lecturer Canan Sümeyra GÜN to conduct this study with me, under the condition that they explain the details clearly and maintain the confidentiality of my personal information. Throughout the study, I pledge not to share the username, password, or application content provided to me with anyone else. I also agree to comply with all the

# FORM 4

rules, to fully cooperate with the researchers, and to contact them immediately if any issue arises. I accept that the results of this study may be used without restriction in publications, reports, or other scientific documents. I also understand that I can withdraw from this study at any time.

Researcher Participant Name-Surname: Title, Name-Surname: Lecturer Canan Sümeyra Gün/Assoc. Prof. Dr. Seher Date: SARIKAYA KARABUDAK Date: Phone No: Phone No: 05458125729/0505 448 37 03 Signature: Signature: Menderes Address: Aydın Adnan

University, Central Campus, Faculty of

Nursing, Aydın 09100